CLINICAL TRIAL: NCT05660005
Title: The Effect of Self Myofascial Release and Stretching Exercises in Individuals With Piriformis Syndrome
Brief Title: Self Myofascial Release in Individuals With Piriformis Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, gizem ergezen, Assistant Professor, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E.10304 / 29.03.2018
Record Dates: First submitted 2022-12-05; First posted 2022-12-21 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Piriformis Muscle Syndrome
Keywords: Piriformis syndrome; Pain; hip; range of motion; sciatica
MeSH Terms: conditions — Piriformis Muscle Syndrome; Pain; Sciatica | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Parallel group study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Piriformis Muscle Stretching (Active Comparator): Stretching based on the FAIR (flexion, adduction and internal rotation) position, which provides the most effective stretching on the piriformis muscle, was demonstrated, and a illustrated brochure containing the explanatory information of the application was given to the group participants. With the ipsilateral hip flexion, adduction and internal rotation, the foot is positioned to the lateral side of the contralateral knee, thus long-term passive stretching is targeted in this position. Individuals were asked to leave a 2-days gap between the two stretching exercise sessions by performing 10 repetitions (minimum duration of 15 s stretching, 30 s rest period between repetitions) 3 sets and 3 days of a week.
  Interventions: Other: Muscle Stretching
- Piriformis Muscle Self Myofascial Release (Active Comparator): The patient was presented with the anatomically localized area of the PiM on a visual anatomy map and they were encouraged to find this area on their body. They were asked to verify the trigger points along the PiM and then sat on the trigger points with the help of a tennis ball. Individuals were taught the PiM-SMR exercise, in which they would make forward-backward, right-left, diagonal and circular movements on the ball using their body weight. There was a continuation of the application with an interval of 2 days; 3 times a day with 10 repetitions (the application was for 1 min and 30s rest period between repetitions).
  Interventions: Other: Self Myofascial Release
- Control Group (Experimental): The individuals who refused to apply stretching or releasing included to the control group. They perform only home exercises of hip strengthening
  Interventions: Other: home exercises

INTERVENTIONS:
Other: Muscle Stretching — Stretching based on the FAIR (flexion, adduction and internal rotation) position, which provides the most effective stretching on the piriformis muscle, was demonstrated, and a illustrated brochure containing the explanatory information of the application was given to the group participants. With the ipsilateral hip flexion, adduction and internal rotation, the foot is positioned to the lateral side of the contralateral knee, thus long-term passive stretching is targeted in this position. Individuals were asked to leave a 2-days gap between the two stretching exercise sessions by performing 10 repetitions (minimum duration of 15 s stretching, 30 s rest period between repetitions) 3 sets and 3 days of a week.
  Other Names: Piriformis Muscle Stretching
  Arms: Piriformis Muscle Stretching
Other: Self Myofascial Release — The patient was presented with the anatomically localized area of the PiM on a visual anatomy map and they were encouraged to find this area on their body. They were asked to verify the trigger points along the PiM and then sat on the trigger points with the help of a tennis ball. Individuals were taught the PiM-SMR exercise, in which they would make forward-backward, right-left, diagonal and circular movements on the ball using their body weight. There was a continuation of the application with an interval of 2 days; 3 times a day with 10 repetitions (the application was for 1 min and 30s rest period between repetitions).
  Arms: Piriformis Muscle Self Myofascial Release
Other: home exercises — The exercise brochure consists of 5 different exercises that include isometric and isotonic strengthening of the hip and surrounding muscles. Isometric contraction of gluteus maximus, hip march, external/internal rotation of hips with theraband, 4 sided straight leg raises were the exercises and prescribed 5 days a week, 10 repetitions, 3 sets. All participants were advised to use analgesics determined by the physician in case of unbearable pain and to apply a hot pack for 10-20 minutes before sessions.
  Arms: Control Group

SUMMARY:
Piriformis syndrome is pain that extends from the hip to the knee, caused by the pressure of the piriformis muscle in the hip on the sciatic nerve. There is no valid protocol for the treatment of this syndrome. Physiotherapists generally use hip strengthening exercises and modalities for pain. In this study, in addition to the classical treatment, we will give two different programs consisting of self-myofascial relaxation and stretching exercises to two different groups for 4 weeks as home exercise. We will question the level of pain that people felt in the hip before starting the exercises and at the 4th week after starting the exercises and measured the hip joint range of motion.

DETAILED DESCRIPTION:
Piriformis syndrome (PS) is a condition caused by compression of the sciatic nerve, causing pain, tingling, and numbness. Although conservative treatment includes hip muscle strengthening and stretching, there is no proven treatment method in the literature.

This study will be conducted to investigate the effect of stretching and myofascial release added to standard physiotherapy treatment in piriformis syndrome.

This prospective, randomized controlled study will be planned to completed with 64 individuals between the ages of 20-40. Participants will be randomized into the Piriformis Muscle Stretch Group (PiM-S) and Piriformis Muscle Self Myofascial Release Group (PiM-SMR). Both groups will be included in a home program of muscle strengthening exercises for 4 weeks. And groups will be subjected to perform stretching and self-myofascial relaxation exercises, respectively, in addition to the home exercise program. The primary outcome of the study is pain intensity, and the secondary outcome is determined as the range of motion (ROM) of the hip.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants
* Aged 20 to 40 years
* Presented leg or hip posterior compartment pain
* Diagnosed with chronic PS and without any other source of pain

Exclusion Criteria:

* Any pathology or acute injury around the hip, sacroiliac joint, or lumbar spine;
* Limb length discrepancy,
* Recent buttock trauma,
* Deep gluteal syndrome,
* Extrapelvic compression of the sciatic nerve or sacral plexus ischiogluteal/ischiofemoral bursitis or impingement, Upper hamstring tendinitis,
* Fibromyalgia, myofascial pain syndrome
* Pregnancy.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2022-05-07 (Actual); Study Completion 2022-12-03 (Actual)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks
  The severity of sciatic pain extending along the hip and leg was questioned with the Visual Analog Scale (VAS). The assessment was based on a horizontal 10 cm scale from 1 (least pain) to 10 (the worst pain ever)

SECONDARY OUTCOMES:
Extension Range of motion of the hip angle | 4 weeks
  Extension ROM was measured while the individual was in the pronee position, the pivot point of the goniometer at the trochanter major, the moving arm aligned on the lateral midline of the femur, and the stable arm aligned parallel to the ground.
Flexion Range of motion of the hip angle | 4 weeks
  Flexion ROM was measured while the individual was in the supine position, the pivot point of the goniometer at the trochanter major, the moving arm aligned on the lateral midline of the femur, and the stable arm aligned parallel to the ground.
Adduction Range of motion of the hip angle | 4 weeks
  Adduction ROM were evaluated in the supine position, with the pivot point on the anterior projection of the trochanter major, the stable arm parallel to the anterior superior of the spina iliaca, and the moving arm on the anterior midline of the femur. Femur approached to the midline
Abduction Range of motion of the hip angle | 4 weeks
  Abduction and adduction ROM were evaluated in the supine position, with the pivot point on the anterior projection of the trochanter major, the stable arm parallel to the anterior superior of the spina iliaca, and the moving arm on the anterior midline of the femur. During the evaluation of abduction, attention was paid to the absence of external rotation of the hip and the absence of internal rotation of the hip in adduction.
External Rotation Range of motion of the hip angle | 4 weeks
  The measurement was taken in a prone position, with the knees flexed to 90°, pivot point on the tibial tubercle, with the stable arm perpendicular to the ground and the mobile arm following the tibial crista. During the evaluation, attention was paid to the absence of hip adduction and abduction movement. Knee turned externally
Internal Rotation Range of motion of the hip angle | 4 weeks
  The measurement was taken in a prone position, with the knees flexed to 90°, pivot point on the tibial tubercle, with the stable arm perpendicular to the ground and the mobile arm following the tibial crista. During the evaluation, attention was paid to the absence of hip adduction and abduction movement. Knee turned internally

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen, PhD, Principal Investigator — Medipol University; Mustafa Sahin, PhD, Study Director — Medipol University
Locations (1):
- Gizem Ergezen, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided